CLINICAL TRIAL: NCT06581991
Title: Valine 50mg/ml and Isoleucine 25mg/ml Oral Solutions for Maple Syrup Urine Disease (MSUD) - Acceptability and Tolerance Study
Brief Title: Liquid Valine and Isoleucine in Maple Syrup Urine Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meta Healthcare Ltd (Industry)
Collaborators: Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVMSUD2022(2)
Record Dates: First submitted 2024-08-13; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Maple Syrup Urine Disease
Keywords: Maple Syrup Urine Disease; MSUD; Valine; Isoleucine
MeSH Terms: conditions — Maple Syrup Urine Disease | interventions — Valine; Isoleucine

STUDY DESIGN:
Intervention Model Description: Prospective, open label, observational study of 5 subjects with MSUD for 56 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Liquid valine and liquid isoleucine administration (Experimental): Liquid valine given for 28 days, liquid isoleucine for 28 days
  Interventions: Dietary Supplement: Valine oral solution (50mg/ml) and isoleucine oral solution (25mg/ml)

INTERVENTIONS:
Dietary Supplement: Valine oral solution (50mg/ml) and isoleucine oral solution (25mg/ml) — Subjects will take valine oral solution (50mg/ml) in place of usual powdered valine supplement for 28 days. Subjects will then take isoleucine oral solution (25mg/ml) in place of their usual powdered isoleucine supplement for 28 days.

SUMMARY:
This is a prospective, observational research study in 5 children with Maple Syrup Urine Disease (MSUD). Subjects who are currently taking a valine and isoleucine supplement for MSUD will be recruited for a 56 day trial, of a new ready-to-use valine supplement and a new ready-to-use isoleucine supplement, to evaluate the tolerability and acceptability of the study products compared with their usual products.

DETAILED DESCRIPTION:
This is a prospective, observational 2-part research study in 5 children with Maple Syrup Urine Disease (MSUD). Subjects who are currently taking a valine and isoleucine supplement for MSUD will be recruited for a 56 day trial, of a new ready-to-use valine supplement (Part 1) and a ready-to-use isoleucine supplement (Part 2), to evaluate the tolerability and acceptability of the study products compared with their usual products.

When an appropriate subject has been identified, they and their parents/ caregivers will be sent a study information sheet via the post. They will be invited to request further information about the study if they wish by contacting the Dietitian. The Dietitian will explain the study in more detail either by telephone or via a face-to-face consultation in a convenient location/preferred venue for the participant and their parent/caregiver. Recruitment of each patient will be by written informed consent, which will be completed by the parents/primary caregivers and taken by the Dietitian. Children will also complete an assent/ consent form. Reimbursement will be offered for any travel expenses incurred for any visits to the hospital that are over and above normal/routine visits.

Subjects will replace their usual daily dose of powdered valine supplement with the equivalent amount of the liquid valine supplement for 28 days (Part 1). They will then return to their usual valine supplement and replace their usual powdered isoleucine supplement with the new liquid isoleucine supplement for a further 28 days (Part 2). The outcome of this assessment will be used in a submission to regulatory authorities to enable the study products to be reimbursable on prescription in the United Kingdom (UK). Subjects will be asked to take the new valine supplement for 28 days (Part 1), then the new isoleucine supplement for 28 days (Part 2). During this time, caregivers will be asked to complete a daily acceptability and tolerance questionnaire recording information on:

* Usage and adherence
* Ease of use and any issues with administration
* Any gastro-intestinal side effects The questions should take a maximum of 10 minutes to complete each day. Additional questions will also be completed at the beginning and end of the study that will consider opinion on both usual valine and isoleucine, and study valine and isoleucine, with respect to taste, appearance, smell, presentation and packaging; ease of administration; how the valine is taken; and any other problems or symptoms.

Weight, height and 3 day dietary intake will also be recorded at the beginning and end of Part 1 and Part 2 of the study. A 3-day food diary will record food/drink intake at the beginning of the study whilst taking their usual supplements (Day -3, -2, -1), for 3 days at the end of Part 1 of the study whilst taking the new valine supplement (Days 26, 27, 28), and for 3 days at the end of Part 2 of the study whilst taking the new isoleucine supplement (Days 54, 55, 56).

Meta healthcare will supply the valine oral solution (50mg/ml) and isoleucine oral solution (25mg/ml) for participants free of charge.

During the 56 day trial, weekly routine blood samples will be posted and analysed for valine, leucine and isoleucine as is usual clinical practice. At recruitment, the previous 4 blood results for valine, leucine and isoleucine will be recorded for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Male and female MSUD patients ≥1 year and <16 years of age.
* Patients diagnosed with MSUD.
* Taking both valine and isoleucine supplements for MSUD and willing to take the new supplements for 56 days.
* Absence of comorbidities.
* Adherence with dietary management and valine and isoleucine supplements.
* Able to understand and comply with the requirements of the investigation and sign the Informed Consent Form/Assent form

Exclusion Criteria:

* Age <1 year old and >16 years old.
* Patients with comorbidities.
* Any moderate to severe acute illness which in the opinion of the Investigator would interfere with the study procedures or study outcome.
* History of poor co-operation, non-adherence with dietary management, or poor adherence to investigation procedures.
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.

Ages: 12 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Daily data on gastrointestinal tolerance | From enrollment to end of treatment at 56 days
  A daily record of any gastrointestinal symptoms compared with usual valine and isoleucine supplement
Acceptability and tolerance | From enrolment to end of treatment at 56
  Qualitative questionnaires at study start and end of Part 1 (28 days) and Part 2 (56 dys) of the study
Daily data on study product adherence | From enrollment to the end of treatment at 56 days
  A daily record of study product intake (actual versus prescribed) to check for adherence
3-day food diaries | From enrollment to the end of treatment at 56 days
  A record of patient food and fluid intake for 3 days to monitor valine intake from food - at enrollment, end of part 1 and end of part 2
Blood results for valine, leucine, isoleucine | From enrollment to end of treatment at 56 days
  Routine weekly blood sample taken at home for valine, leucine and isoleucine and posted to the hospital. These will be compared with blood results prior to study commencement to check for any changes

SECONDARY OUTCOMES:
Weight and height measurement | From enrollment to the end of treatment at 56 days
  Weight and height will be measured at enrollment, end of Part 1 (28 days) and end of Part 2 (56 days) of the study to check that growth is adequate

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Principal Investigator — Birmingham Children's Hospital, UK

IPD SHARING:
Plan to Share IPD: No
No identifiable individual patient data will disclosed outside of the clinical care team.